CLINICAL TRIAL: NCT05215912
Title: A Phase 1, Double-blind, Single- and Multiple-ascending Dose Escalation Study of TNB-738, a Biparatopic Antibody Targeting CD38 in Healthy Volunteers
Brief Title: A Single and Multiple Dosing Study Targeting Biparatopic Antibody CD38 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TeneoFour Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Organization: Ancora Biotech LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNB-738
Record Dates: First submitted 2021-11-23; First posted 2022-01-31 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteer
Keywords: CD38

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single Ascending Dose (SAD -Arm A) (Experimental): Up to 5 cohorts of subjects receiving sequentially ascending dose of TNB-738 or placebo are planned until maximum tolerated dose is reached or recommended phase 2 dose is identified
  Interventions: Drug: TNB-738
- Multiple Ascending Dose (MAD- Arm B) (Experimental): An expansion cohort (upto 4 cohorts) will be enrolled after maximum tolerated dose or recommended phase 2 dose is established.
  Interventions: Drug: TNB-738

INTERVENTIONS:
Drug: TNB-738 — TNB-738 is an investigation drug. Other: Matching placebo
  Arms: Single Ascending Dose (SAD -Arm A)
Drug: TNB-738 — TNB-738 is an investigation drug. Other: Matching placebo
  Arms: Multiple Ascending Dose (MAD- Arm B)

SUMMARY:
This is a Phase 1, Double blind, Single ascending and Multiple ascending dose (SAD and MAD) escalation study in Healthy Volunteers.

DETAILED DESCRIPTION:
TNB-738 is a fully human bispecific antibody used to inhibit human CD38 enzyme.

The study will consist of 2 arms (A and B). The SAD arm (Arm A) of the study consists of sequential single dose escalation cohorts, whereas the MAD portion (Arm B) of the study consists of sequential dose escalation cohorts receiving study drug once every 4 weeks for 3 doses. In both Arm A and Arm B, subjects will be randomized to receive either TNB-738 or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female
2. Age 18 - 75
3. Body mass index (BMI) ranging between 18 and 35 kg/m2, inclusive
4. Female subjects of child-bearing potential must agree to use one of the study-approved effective contraceptive methods for the duration of the study
5. Male subjects must practice true abstinence or agree to use a condom while participating in the study through End of study (EOS)
6. If female, a negative serum pregnancy test at Screening and urinary pregnancy test at Day -1 is required
7. Able to read, understand, and provide signed informed consent
8. Able to communicate adequately with the investigator and to comply with the requirements for the entire study.

Exclusion Criteria:

1. Subject has any significant medical condition that would prevent the subject from participating in the study.
2. Subject is pregnant or breastfeeding.
3. Subject is currently receiving treatment with a biologic agent.
4. Subject has a history of anaphylactic reactions to biologic agents.
5. Subject has been dosed with another investigational drug study within 60 days prior to study drug administration.
6. Subject has current or recent (within 4 weeks prior to screening) signs or symptoms of infection that require antibiotic administration.
7. Subject has evidence of COVID-19 infection and/or subject is deemed at risk for the coronavirus disease in the opinion of the investigator or the subject has participated in another clinical study involving treatment(s), which may increase such risk.
8. Subject has used any prescription (excluding hormonal birth control) drugs within 14 days or illicit drugs within 30 days, or 5 half-lives (whichever is longer), prior to study drug administration.
9. Subject has a positive urine drug test or alcohol breath test at screening.
10. Subject has donated or lost more than 1 unit of blood (500 mL) within 60 days or more than 1 unit of serum within 7 days before the study drug administration.
11. Subject is HIV, HBV, or HCV positive.
12. Subject has received a live virus vaccine within 4 weeks of dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of TNB-738 by the incidence of treatment emergent adverse events in Single Ascending group. Adverse Events will be graded according to the NCI-CTCAE, version 5.0 | 13 weeks
Safety and tolerability of TNB-738 by the incidence of treatment emergent adverse events in Multiple Ascending group. Adverse Events will be graded according to the NCI-CTCAE, version 5.0 | 21 weeks
To investigate the Cmax (maximum Serum concentration) of TNB-738 following Single Ascending Dose. | 13 weeks
To investigate the Cmax (Maximum Serum concentration) of TNB-738 following Multiple Ascending Dose | 21 weeks
Tmax (time for maximum serum concentration) for Single Ascending Dose | 13 weeks
Tmax (time for maximum serum concentration) for Multiple Ascending Dose | 21 weeks
Terminal elimination half-life (t1/2) for Single Ascending Dose | 13 weeks
Terminal elimination half-life (t1/2) for Multiple Ascending Dose | 21 weeks

SECONDARY OUTCOMES:
Anti drug antibodies (ADA) as a measurement of immunogenicity following Single Ascending Dose of TNB-738 | 13 weeks
Anti drug antibodies (ADA) as a measurement of immunogenicity following Multiple Ascending Dose of TNB-738 | 21 weeks
To determine CD38 enzyme activity following Single Ascending Dose | 13 weeks
To determine CD38 enzyme activity following Multiple Ascending Dose | 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ben Buelow, MD, PhD, Study Director — TeneoFour Inc.
Locations (1):
- Q-Pharm Pty Ltd, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No